CLINICAL TRIAL: NCT05506033
Title: Optimization of Glucocorticoid Taper Strategies for Maintenance Therapy of Systemic Lupus Erythematosus Associated Immune Thrombocytopenia (SLE-ITP)
Brief Title: Optimization of Glucocorticoid Taper Strategies for SLE-ITP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tanklhj@163.com
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-07

CONDITIONS: Lupus Erythematosus, Systemic; Purpura, Thrombocytopenic, Idiopathic; Glucocorticoids; Adverse Effect of Glucocorticoids
Keywords: GCs taper strategy; Lupus Erythematosus, Systemic; Purpura, Thrombocytopenic, Idiopathic
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard GCs taper group (No Intervention): After a complete response (PLT ≥100x10^9/L) was confirmed, the dose of prednisone (or equivalent dose of glucocorticoids) would be reduced by 2 tablets every two weeks. When it reaches 6 tablets /d, the dose would be reduced by 1 tablet every 2 weeks, and when it reaches 15mg/d, the dose would be reduced by half tablet every 2 weeks.
- rapid GCs taper group (Experimental): After a complete response (PLT ≥100x10^9/L) was confirmed, the dose of prednisone (or equivalent dose of glucocorticoids) would be cut in half (25mg/d for weight less than 50kg, 30mg/d for weight 50-75kg , 40mg/d for weight more than 75kg ). After that, the dose would be reduced by 2 tablets every two weeks. When it reaches 6 tablets /d, the dose would be reduced by 1 tablet every 2 weeks, and when it reaches 15mg/d, the dose would be reduced by half tablet every 2 weeks.
  Interventions: Procedure: rapid GCs taper

INTERVENTIONS:
Procedure: rapid GCs taper — After a complete response was achieved, the GCs dose was halved from the original dose.
  Arms: rapid GCs taper group

SUMMARY:
SLE associated immune thrombocytopenia (SLE-ITP) is one of the main clinical manifestations of SLE. Approximately 70% of SLE patients follow a relapsing-remitting course. Similarly, SLE-ITP often relapses during GCs tapering. At the same time, patients with SLE-ITP may suffer from thrombocytopenia and damage to vital organs when they relapse, seriously affecting their lives. Therefore, maintenance therapy after remission is an inevitable choice for SLE-ITP.

The SLE guidelines recommend GCs and immunosuppressive agents(ISA) are first-line maintenance treatment in the treatment of SLE-ITP. GCs is indispensable in SLE treatment, but it is associated with a series of side effects, which are related to the dosage and duration of use. How to maintain remission with the most appropriate dose of GCs is a problem that needs to be considered in clinical practice. However, the existing guidelines lack detailed recommendations on the specific use of GCs in maintenance therapy for SLE-ITP, and there is also a lack of relevant clinical studies to guide. The GCs reduction regimen commonly used in maintenance therapy is a gradual reduction after 1 month of adequate GCs therapy, usually by 10% of the original dose every 2 weeks. However, the side effects of this reduction method are obvious, and whether the treatment can be maintained with less cumulative dose and maintenance duration of GCs is an urgent problem to be solved.

Clinical observations show that in a small number of patients with relative contraindications to GCs, a more rapid taper can maintain an effective response. Currently, rapid dosing reduction is recommended in both Lupus nephritis(LN) and the ANCA-associated nephritis guidelines of ACR. However, SLE-ITP changes more rapidly than LN. Although similar maintenance responses have been observed in a few patients between rapid dosing reduction and conventional method, relevant clinical studies are lacking. It is necessary to explore the effectiveness of rapid GCs tapering method.

Therefore, the investigators plan to conduct a single-center, prospective, randomized design, non-blind, non-inferiority controlled study on the optimization of GCs taper strategy for SLE-ITP maintenance therapy.In this study,sustained response rate and relapse rate within 3 months and 6 months were observed to judge the effectiveness of rapid GCs taper strategy, thus providing a basis for clinical GCs taper strategy.

DETAILED DESCRIPTION:
Complete response was defined as a platelet count ≥100x10^9/L and the absence of bleeding and new other symptoms.Complete response would be confirmed by platelet counts on 2 separate occasions 7 days apart. Adequate glucocorticoids treatment was defined as at least a dose 50mg/day of prednisone (or equivalent glucocorticoids) for patients with weight less than 50kg, 60mg/day for patients with weight 50-75kg , 75mg/day for patients with weight more than 75kg. Adequate glucocorticoids were used for induction, and the total duration of adequate glucocorticoids treatment for patients enrolled was no longer than 3 weeks.Neither Thrombopoietin receptor agonist(TPO-RA) nor intravenous immunoglobulin(IVIG)were permitted in induction therapy or maintenance therapy.In addition to hydroxychloroquine(HCQ), other immunosuppressive agents are not permitted in induction therapy or maintenance therapy. After confirmation of complete response, the patients enrolled were randomly divided into two groups according to two different methods of GCs taper.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 14-75 (including 14 and 75);
2. It meets the 2012 Systemic lupus Erythematosus International Collaborative Group (SLICC) classification criteria or the 2019 ACR and European Society of Rheumatology (EULAR) classification criteria ;
3. severe SLE-ITP patients with PLT≤30x10^9/L at onset and complete response (PLT ≥100x10^9/L) after induction therapy within 3 weeks;
4. Prior to the commencement of any study-specific procedure, the patient or legal representative must provide signed and dated written informed consent.

Exclusion Criteria:

1. Relapse in the presence of glucocorticoid and/or immunosuppressive maintenance therapy;
2. Combined with antiphospholipid syndrome;
3. Combined with other important organ damage such as lupus nephritis, neuropsychiatric lupus;
4. Coexisting immune diseases require glucocorticoid and/or immunosuppressive therapy;
5. There are serious comorbidities affecting treatment such as diabetes, severe hypertension, coronary heart disease;
6. self-evaluation affected by poor understanding ability, vision decline and other reasons ;
7. Poor adherence and failure to adhere to treatment as prescribed. -

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
significant relapse | within 12 weeks
  significant relapse were defined as 1 or more of the following: 1)a platelet count<30x10^9/L or less than 2-fold increase of the baseline platelet count or bleeding;2)new damage to important organs(renal, central nervous system, cardiopulmonary, vasculitis, myositis,fever, active hemolytic anemia or gastrointestinal activity);3)manifestations requiring an increase in prednisone(or equivalent) to >0.5mg/kg/day;4)SLEDAI-2K instrument score greater than 12;5) change in physician's global assessment score from baseline to greater than 2.5.
significant relapse | within 24 weeks
  significant relapse were defined as 1 or more of the following: 1)a platelet count<30x10^9/L or less than 2-fold increase of the baseline platelet count or bleeding;2)new damage to important organs(renal, central nervous system, cardiopulmonary, vasculitis, myositis,fever, active hemolytic anemia or gastrointestinal activity);3)manifestations requiring an increase in prednisone(or equivalent) to >0.5mg/kg/day;4)SLEDAI-2K instrument score greater than 12;5) change in physician's global assessment score from baseline to greater than 2.5.

SECONDARY OUTCOMES:
Mild to moderate relapse | within 12 weeks
  Mild to moderate relapse were defined as 1 or more of the following: 1)30x10^9/L≤ a platelet count <100x10^9/L and at least 2-fold increase of the baseline count and absence of bleeding and new damage to important organs（renal, central nervous system, cardiopulmonary, vasculitis, fever, active hemolytic anemia or gastrointestinal activity);2)any manifestations requiring an increase in prednisone(or equivalent) not greater than 0.5mg/kg/day;3)greater than 3-point change in SLEDAI-2K instrument score, with total score of 12 or less;4)or change in the physician's global assessment score of 1.0 or more but remaining 2.5 or less.
Mild to moderate relapse | within 24 weeks
  Mild to moderate relapse were defined as 1 or more of the following: 1)30x10^9/L≤ a platelet count <100x10^9/L and at least 2-fold increase of the baseline count and absence of bleeding and new damage to important organs（renal, central nervous system, cardiopulmonary, vasculitis, fever, active hemolytic anemia or gastrointestinal activity);2)any manifestations requiring an increase in prednisone(or equivalent) not greater than 0.5mg/kg/day;3)greater than 3-point change in SLEDAI-2K instrument score, with total score of 12 or less;4)or change in the physician's global assessment score of 1.0 or more but remaining 2.5 or less.
Clinical remission | at 24 weeks
  According to DORIS's definition of SLE remission in 2021.
a Lupus Low Disease Activity State | at 24 weeks
  According to the definition of SLE low disease activity state formulated in 2015.

CONTACTS AND LOCATIONS:
Overall Officials: He-Jun Li, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanouriakis A, Kostopoulou M, Alunno A, Aringer M, Bajema I, Boletis JN, Cervera R, Doria A, Gordon C, Govoni M, Houssiau F, Jayne D, Kouloumas M, Kuhn A, Larsen JL, Lerstrom K, Moroni G, Mosca M, Schneider M, Smolen JS, Svenungsson E, Tesar V, Tincani A, Troldborg A, van Vollenhoven R, Wenzel J, Bertsias G, Boumpas DT. 2019 update of the EULAR recommendations for the management of systemic lupus erythematosus. Ann Rheum Dis. 2019 Jun;78(6):736-745. doi: 10.1136/annrheumdis-2019-215089. Epub 2019 Mar 29. PMID 30926722
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Chung SA, Langford CA, Maz M, Abril A, Gorelik M, Guyatt G, Archer AM, Conn DL, Full KA, Grayson PC, Ibarra MF, Imundo LF, Kim S, Merkel PA, Rhee RL, Seo P, Stone JH, Sule S, Sundel RP, Vitobaldi OI, Warner A, Byram K, Dua AB, Husainat N, James KE, Kalot MA, Lin YC, Springer JM, Turgunbaev M, Villa-Forte A, Turner AS, Mustafa RA. 2021 American College of Rheumatology/Vasculitis Foundation Guideline for the Management of Antineutrophil Cytoplasmic Antibody-Associated Vasculitis. Arthritis Rheumatol. 2021 Aug;73(8):1366-1383. doi: 10.1002/art.41773. Epub 2021 Jul 8. PMID 34235894
- [Result] Fanouriakis A, Tziolos N, Bertsias G, Boumpas DT. Update omicronn the diagnosis and management of systemic lupus erythematosus. Ann Rheum Dis. 2021 Jan;80(1):14-25. doi: 10.1136/annrheumdis-2020-218272. Epub 2020 Oct 13. PMID 33051219
- [Result] Jung JH, Soh MS, Ahn YH, Um YJ, Jung JY, Suh CH, Kim HA. Thrombocytopenia in Systemic Lupus Erythematosus: Clinical Manifestations, Treatment, and Prognosis in 230 Patients. Medicine (Baltimore). 2016 Feb;95(6):e2818. doi: 10.1097/MD.0000000000002818. PMID 26871854
- [Result] Chinese Rheumatology Association; National Clinical Research Center for Dermatologic and Immunologic Diseases; Chinese Systemic Lupus Erythematosus Treatment and Research Group. [2020 Chinese guidelines for the diagnosis and treatment of systemic lupus erythematosus]. Zhonghua Nei Ke Za Zhi. 2020 Mar 1;59(3):172-185. doi: 10.3760/cma.j.issn.0578-1426.2020.03.002. Chinese. PMID 32146743